CLINICAL TRIAL: NCT05365711
Title: Carriage of Beta Haemolytic Streptococci During Pregnancy
Status: Active, not recruiting | Type: Observational
Sponsor: Turku University Hospital (Other Government)
Collaborators: University of Turku (Other)
Responsible Party: Sponsor
Other Study IDs: 67/1801/2021
Record Dates: First submitted 2022-04-26; First posted 2022-05-09 (Actual); Last update posted 2024-03-21 (Actual); Status verified 2024-03

CONDITIONS: Pregnancy Related
Keywords: pregnancy; group a streptococci; group b streptococci; carriage; microbiota; Streptococcus pyogenes; Streptococcus agalactiae

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Biospecimen Retention: Samples Without DNA — saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnant women: Microbiological samples are collected from the pregnant women in the mid-pregnancy and during the delivery. Patient records of these women and newborns are investigated for any infections or complications during and after the delivery.
- Partners: Partners of the pregnant women will be studied to understand the household transmission of studied bacteria and possible risk factors for carriage.

SUMMARY:
This is a prospective clinical study that aims to investigate asymptomatic carriage of beta haemolytic streptococci (especially group A streptococci, GAS and group B streptococci, GBS) during pregnancy. Association of asymptomatic carriage to possible complications of the mother or the newborn as well as the transmission between spouses will be evaluated. Maternal microbiota during labour will also be studied.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women
* partner of the pregnant women
* over/equal 18 years of age
* willing to participate the study

Exclusion Criteria:

* multiple pregnancy
* age <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women and their partners
Study Population: Pregnant women attending ultrasound scan are asked to participate in the study. Partners of the pregnant women are asked to participate as well.
Sampling Method: Non-Probability Sample
Enrollment: 1040 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Carriage of beta haemolytic streptococci | up to 30 weeks
  Throat and vaginal carriage of beta haemolytic streptococci (especially GAS and GBS) during pregnancy. Transmission and longitude of the carriage will be evaluated as well.

SECONDARY OUTCOMES:
Pregnancy or delivery related infections/complications | up to12 weeks
  Patient records of the pregnant women will be surveyed for any complications/infections until 12 week after delivery. Data will be analysed together with the microbiological findings from the women.
Infections/complications of newborn | 12 weeks after birth
  Patient records are surveyed to search for any infections/complications of the newborn until 12 weeks of age. Data will be analysed together with the findings from their mother.

CONTACTS AND LOCATIONS:
Locations (1):
- Turku University Hospital, Turku, Finland